CLINICAL TRIAL: NCT06598982
Title: Investigation of Respiratory Muscle Sarcopenia in Patients with Systemic Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin GEDIKLI, Faculty of Health Sciences Physiotherapy and Rehabilitation-Research assistant, Selcuk University
Other Study IDs: SelcukU-FTR-YG-02
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Sclerosis (SSc); Scleroderma
Keywords: respiration; sarcopenia; diaphragm; muscle strength
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Respiratory Aspiration; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with systemic sclerosis

SUMMARY:
The aim of this study was to investigate respiratory muscle sarcopenia in individuals with systemic sclerosis. The main question it aims to answer is:

What is the prevalence of respiratory muscle sarcopenia in patients with systemic sclerosis? Participants body composition (bioelectrical impedance), hand grip strength (hand dynanometer), physical performance tests (5 repetition sit-and-stand test, 4-meter walk test, Timed up-and-go test) and respiratory muscle strength were evaluated.

DETAILED DESCRIPTION:
Sarcopenia is a generalized and progressive loss of skeletal muscles and is characterized by a decrease in muscle strength, muscle mass and physical performance. It usually occurs in older people, but can also occur in people with certain diseases or who lead a very sedentary lifestyle. The European Working Group on Sarcopenia in Older People (EWGSOP) has developed guidelines for diagnosing sarcopenia and determining its severity. EWGSOP defined three conceptual stages of sarcopenia. Pre-sarcopenia is characterized by low muscle mass that does not affect muscle strength or physical performance. Sarcopenia is characterized by low muscle mass and decreased muscle strength or reduced physical performance. Severe sarcopenia is characterized when all criteria are met. Respiratory muscle sarcopenia is defined as a condition of muscle fiber atrophy and weakness that also occurs in respiratory muscles. The Japanese Respiratory Sarcopenia Study Group defined respiratory muscle sarcopenia as "whole body sarcopenia and low respiratory muscle mass with low respiratory muscle strength and/or low respiratory function". Respiratory muscle sarcopenia was also defined by Kera et al. based on peak expiratory flow rate. However, whole body sarcopenia and respiratory muscle strength are also important to define and diagnose respiratory muscle sarcopenia. The incidence of respiratory muscle sarcopenia is higher in the presence of sarcopenia. Sarcopenic respiratory failure is diagnosed when there is sarcopenia with functional impairment. Cases of respiratory sarcopenia without functional impairment are diagnosed as "at risk of sarcopenic respiratory failure". When the literature is reviewed, it is seen that there is no study on respiratory muscle sarcopenia in patients with systemic sclerosis. Therefore, the aim of this study is to examine respiratory muscle sarcopenia in patients with systemic sclerosis.

The smallest sample size of the study was 85 people with 90% power at 95% confidence interval. Data will be analyzed using IBM® SPSS® Statistics for Windows (ver. 25.0; IBM Corp, New York, USA) software. Values will be expressed as mean ± standard deviation and median (25-75 quartiles) for continuous variables and frequencies will be reported for categorical variables. Shapiro-Wilk test and histograms will be used to assess the normality distribution of the data. Pearson correlation coefficient will be used to evaluate the parameters associated with respiratory muscle strength. Binary Logistic Regression Analysis, which is used to estimate whether the dependent variable belongs to two categorical classes, will be used to determine the risk factors for respiratory muscle sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* 2013 To be diagnosed with systemic sclerosis according to ACR/EULAR classification criteria
* Being clinically stable
* Ability to adapt to tests (visual, cognitive, cooperative)

Exclusion Criteria:

* Those with neurological and/or musculoskeletal problems that may affect the work
* Presence of severe joint contracture or painful ulcers that may affect muscle strength measurement and walking
* Presence of severe infection or sepsis
* Being diagnosed with a known additional rheumatologic disease
* Any stage of cancer
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Selçuk University, Faculty of Health Sciences. The study will include volunteer individuals with systemic sclerosis who are eligible to participate in the study and who are being followed up and treated with a diagnosis of scleroderma in the Department of Rheumatology.
  -- Purposive sampling
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Sarcopenia Assessment | baseline
  The diagnosis of respiratory muscle sarcopenia will also be made by combining the results of secondary measurements.
  Participants included in the study:
  * Hand grip strength <27 kg for men and <16 kg for women,
  * Bioelectrical Impedance Analysis (Skeletal muscle mass (SMM)<20 kg for men and < 15 kg for women) the participant is diagnosed with sarcopenia. They will also be diagnosed with a frailty phenotype based on the results of the Timed Stand and Walk Test, the 4 meter walk test and the 5 Repetition Sit and Stand Test.
  Patients diagnosed with sarcopenia will be diagnosed with respiratory muscle sarcopenia if respiratory muscle weakness is also detected.

SECONDARY OUTCOMES:
Grip Force Measurement | baseline
  The hand muscle grip strength of the individuals will be measured with a hand dynamometer. During the measurement, the position recommended by the American Association of Hand Therapists (ASHT); the participant will be in an upright sitting position and no arm support will be allowed on the sitting surface. The elbow and knee angle will be set to 90°. The wrist will be held without deviation. The measurement will be performed 3 times with an interval of 10 seconds and the highest value will be used in the study.
4 Meter Walking Speed Test (4MWT) | baseline
  4MWT is a measure of walking speed, a vital sign of mobility and functionality. In older adults, walking speed is a clinical indicator of conditions such as frailty and sarcopenia. Participants were instructed to start walking at their normal speed 2 m behind the "start point" and continue until they passed the "end point". Using a stopwatch, the time taken for each participant to walk the 4 m distance between the "start" and "end" point will be measured. This will be used to calculate walking speed (distance/time).
Timed Up and Go Test (TUG) | baseline
  This functional test measures the time it takes for an individual to stand up from a standard chair, walk 3 m at normal speed, turn around, walk back to the starting point and sit down. Using a stopwatch, participants test scores are recorded in seconds.
5 Repetition Sit and Stand Test | baseline
  An armless chair with a straight back support and a rigid seat at a height of 48 cm from the floor will be fixed to the wall. Participants will be asked to sit on the chair and come forward in the chair until their feet are flat on the floor. Participants will be asked to do a "stand and sit" movement once with their arms crossed across their chest. The test will be terminated for those who cannot complete the task or need assistance. Those who successfully complete the first task will be asked to perform five consecutive stand and sit as fast as possible. The timing is started with the command start and stopped at the end of the fifth posture. Our participants test scores will be recorded in seconds using a stopwatch.
Respiratory muscle strength | baseline
  Intraoral pressure will be measured with a measuring device. They are easily applicable and simple measurements. Maximal voluntary inspiratory and expiratory pressures (MIP and MEP) are the most commonly used noninvasive methods to measure respiratory muscle strength. It is based on Müller (maximal inspiration) and Valsalva (maximal expiration).
Demographic and Clinical Information | baseline
  Information on age, height (meter), body weight (kg), body mass index(kg/m²), gender, educational status, occupation, medication use, exercise habits and disease will be evaluated. These data will be recorded on pre-prepared forms.
Body composition | baseline
  Body mass and body composition will be measured using bioelectrical impedance method. The variables to be assessed are body mass index (BMI = body mass (kg)/height2 (m)2 ), fat mass (pFM) expressed as a percentage of body mass, fat-free mass (FFM) expressed in kilograms, and appendicular skeletal muscle mass (ASMM) and skeletal muscle mass (SMM) expressed in kilograms. Data will be collected with a bioelectrical impedance device and recorded on pre-prepared forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sousa-Santos AR, Amaral TF. Differences in handgrip strength protocols to identify sarcopenia and frailty - a systematic review. BMC Geriatr. 2017 Oct 16;17(1):238. doi: 10.1186/s12877-017-0625-y. PMID 29037155
- [Background] Nagano A, Wakabayashi H, Maeda K, Kokura Y, Miyazaki S, Mori T, Fujiwara D. Respiratory Sarcopenia and Sarcopenic Respiratory Disability: Concepts, Diagnosis, and Treatment. J Nutr Health Aging. 2021;25(4):507-515. doi: 10.1007/s12603-021-1587-5. PMID 33786569
- [Background] Mehmet H, Robinson SR, Yang AWH. Assessment of Gait Speed in Older Adults. J Geriatr Phys Ther. 2020 Jan/Mar;43(1):42-52. doi: 10.1519/JPT.0000000000000224. PMID 30720555
- [Background] Maggio M, Ceda GP, Ticinesi A, De Vita F, Gelmini G, Costantino C, Meschi T, Kressig RW, Cesari M, Fabi M, Lauretani F. Instrumental and Non-Instrumental Evaluation of 4-Meter Walking Speed in Older Individuals. PLoS One. 2016 Apr 14;11(4):e0153583. doi: 10.1371/journal.pone.0153583. eCollection 2016. PMID 27077744
- [Background] Kera T, Kawai H, Hirano H, Kojima M, Watanabe Y, Motokawa K, Fujiwara Y, Ihara K, Kim H, Obuchi S. Definition of Respiratory Sarcopenia With Peak Expiratory Flow Rate. J Am Med Dir Assoc. 2019 Aug;20(8):1021-1025. doi: 10.1016/j.jamda.2018.12.013. Epub 2019 Feb 6. PMID 30737167
- [Background] Hulzebos E, Takken T, Reijneveld EA, Mulder MMG, Bongers BC. Reference Values for Respiratory Muscle Strength in Children and Adolescents. Respiration. 2018;95(4):235-243. doi: 10.1159/000485464. Epub 2018 Jan 17. PMID 29342462
- [Background] Greco F, Tarsitano MG, Cosco LF, Quinzi F, Folino K, Spadafora M, Afzal M, Segura-Garcia C, Maurotti S, Pujia R, Pujia A, Buono P, Emerenziani GP. The Effects of Online Home-Based Pilates Combined with Diet on Body Composition in Women Affected by Obesity: A Preliminary Study. Nutrients. 2024 Mar 21;16(6):902. doi: 10.3390/nu16060902. PMID 38542813
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Cesari M, Kritchevsky SB, Newman AB, Simonsick EM, Harris TB, Penninx BW, Brach JS, Tylavsky FA, Satterfield S, Bauer DC, Rubin SM, Visser M, Pahor M; Health, Aging and Body Composition Study. Added value of physical performance measures in predicting adverse health-related events: results from the Health, Aging And Body Composition Study. J Am Geriatr Soc. 2009 Feb;57(2):251-9. doi: 10.1111/j.1532-5415.2008.02126.x. PMID 19207142
- [Background] Calderon LM, Pope JE. Scleroderma epidemiology update. Curr Opin Rheumatol. 2021 Mar 1;33(2):122-127. doi: 10.1097/BOR.0000000000000785. PMID 33481429